CLINICAL TRIAL: NCT03839745
Title: Short-Term Cardiovascular Effects of E-Cigarettes: Influence of Device Power
Acronym: TCORS-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1723965; 5U54HL147127 (NIH); NCI-2021-01564 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2019-01-24; First posted 2019-02-15 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Risk Factor; Nicotine Dependence
Keywords: E-Cigarettes; Vaping; E-Cig Mods
MeSH Terms: conditions — Tobacco Use Disorder; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Power level 10, 15, or 20 watts (Other): Using an electronic cigarette, the patient will participate in a standardized vaping session using 1 of 3 assigned battery power levels
  Interventions: Other: Electronic Cigarette
- 1 of the other 2 remaining power levels (Other): Using an electronic cigarette, the patient will participate in a standardized vaping session using 1 of the other 2 remaining power levels
  Interventions: Other: Electronic Cigarette
- Remaining power level (Other): Using an electronic cigarette, the patient will participate in a standardized vaping session using the remaining power level
  Interventions: Other: Electronic Cigarette

INTERVENTIONS:
Other: Electronic Cigarette — E-cigarette Device: The delivery device will be a variable wattage all-in-one device with operating wattage of 7.0 - 75.0 W, which is inclusive of the three power levels we intend to study.

SUMMARY:
This study will examine the short-term cardiovascular (CV) effects of e-cigarette device power in a randomized, crossover clinical and behavioral pharmacology study of experienced adult e-cigarette users (N=21). The specific aim is to determine the impact of e-cigarette power on nicotine pharmacology, systemic exposure to toxic volatile organic compounds (VOCs), and short-term cardiovascular effects.

DETAILED DESCRIPTION:
This is a single-site, randomized, crossover study of experienced adult e-cigarette users to assess nicotine exposure, toxicant exposure, and the short-term CV effects of e-cigarette power. Three power levels will be assessed on all participants: 10, 15, and 20 watts.

Hypothesis 1a: Systemic nicotine exposure and subjective measures of sensation in the throat, reward, and satisfaction will increase with increasing power in the e-cigarette device.

Hypothesis 1b: Mercapturic acid metabolites of volatile organic compounds (VOCs), particularly acrolein, will increase with e-cigarette power.

Hypothesis 1c: CV effects increase with higher power, and are manifested as changes in hemodynamic parameters, hormonal release, and biomarkers of endothelial function, platelet activation, inflammation, and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Use e-cigarettes on at least 25 days in the past 30 for at least 3 months and have not used another tobacco product in the past 30 days
* Healthy on the basis of medical history and limited physical examination (screening visit), as described below:
* Heart rate < 105 beats per minute (BPM)*
* Systolic Blood Pressure < 160 and > 90*
* Diastolic Blood Pressure < 100 and > 50*
* Body Mass Index (BMI) ≤ 38.0 (at investigator's discretion for higher BMI if no other concurrent health issues)

  *Considered out of range if both machine and manual readings are above/below these thresholds.
* Any race/ethnicity

Exclusion Criteria:

* Used tobacco products other than e-cigarettes in past 30 days
* Expired carbon monoxide of over 5 ppm at screening
* The following unstable medical conditions:
* Heart disease
* Uncontrolled hypertension
* Thyroid disease (not hypo or hyper, controlled with medication)
* Diabetes
* Hepatitis B or C or Liver disease
* Glaucoma
* Prostatic hypertrophy
* Psychiatric conditions:
* Current or past schizophrenia, and/or current or past bipolar disorder
* Adult onset attention deficit hyperactivity disorder (ADHD) (if being treated)
* Participants with current or past depression and/or anxiety disorders will be reviewed by the study physician and considered for inclusion
* Psychiatric hospitalizations are not exclusionary, but study participation will be determined as per study physician's approval
* Drug/Alcohol Dependence:
* Alcohol or illicit drug dependence within the past 12 months with the exception of those who have recently completed an alcohol/drug treatment program
* Positive toxicology test at the screening visit (THC & prescribed medications okay)
* Opioid replacement therapy
* Positive urine cannabis is not exclusionary but participant must report use of cannabis in any form on not more than 2 times per week to be eligible
* Psychiatric medications:
* Current regular use of any psychiatric medications with the exception of Selective Serotonin Reuptake Inhibitor (SSRI) and serotonin-norepinephrine reuptake Inhibitor (SNRIs) and current evaluation by the study physician that the participant is otherwise healthy, stable, and able to participate.
* Medications
* Use of medications that are inducers of nicotine metabolizing enzyme CYP2A6 (Example: rifampicin, dexamethasone, phenobarbital, and other anticonvulsant drugs).
* Concurrent use of nicotine-containing medications
* Other/Misc. Chronic Health Conditions
* Oral thrush
* Fainting
* Untreated thyroid disease
* Other "life threatening illnesses" as per study physician's discretion
* Pregnancy
* Pregnancy (self-reported and urine pregnancy test)
* Breastfeeding (determined by self-report)
* Concurrent participation in another clinical trial
* Inability to communicate in English
* Planning to quit smoking or vaping within the next 60 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mean nicotine levels | Day 1 of each Arm
  Concentration of plasma nicotine (ng/ml) will be used to assess differences in nicotine exposure across the three power levels.
Mean scores on the Minnesota Nicotine Withdrawal Scale (MNWS) | Days 1-2 of each Arm
  The Minnesota Nicotine Withdrawal Scale (MNWS) is an 7-item self-report scale designed to measure the severity of craving and withdrawal symptoms experienced during smoking cessation. Each item is rated on a scale of 0 to 4 with 0=none,1= Slight, 2= Mild, 3= Moderate, and 4=Severe. Seven of the items are symptoms derived from the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) Tobacco Withdrawal diagnosis and are as follows: depression, insomnia, irritability/frustration/anger, anxiety/nervousness, difficulty concentrating, restlessness, increased appetite and at least five of the items must have responses in order to generate a reliable score. Responses to each item are summed to produce a total withdrawal summary score. The overall mean and standard deviation (SD) will be calculated with a minimum score of 0 and a maximum mean score of 28. Greater scores indicate a higher level of severity in withdrawal symptoms.
Mean scores on the Questionnaire of Smoking Urges (QSU-Brief) | Days 1-2 of each Arm
  The QSU-Brief consists of 10 statements about the respondent's feelings and thoughts about participant's desire to smoke cigarettes as the participant is completing the questionnaire (i.e., right now). Each response is scored a number ranging from 1 (strongly disagree) to 7 (strongly agree) and scores are calculated by summing the item scores for a total score where a higher scores (score range from 10 points to 70 points) indicates a higher intensity of the indicated subjective effect.
Mean scores on the modified Cigarette Evaluation Scale (mCES) | Days 1-2 of each Arm
  We will compile a score for the subjective effect of reward using the sum of points scored in the five subscales (Smoking Satisfaction - score range from 1 point to 7 points; Psychological Reward - score range from 5 points to 35 points; Aversion - score range from 2 points to 14 points; Enjoyment of Respiratory Tract Sensations - score range from 2 points to 14 points; and Craving Reduction - score range from 1 point to 7 points) of the modified Cigarette Evaluation Scale (mCES), where a higher score indicates a higher intensity of the indicated subjective effect.
Mean differences in acrolein (3HPMA) | Day 2 of each Arm
  Mean differences in 24-hour urine mercapturic acid metabolites of VOCs, particularly 3HPMA, the metabolite of acrolein across power settings will be calculated to determine Volatile Organic Compounds (VOC) Exposure.
Mean Heart Rate | Days 1-3 of each Arm
  Heart rate for participants will be measured in beats per minute throughout the inpatient stay as a measure of cardiovascular effects.
Mean Blood Pressure | Day 2 of each Arm
  Participant systolic and diastolic blood pressure for participants will be taken for 24 hours during ad-lib e-cigarette use as a measure of cardiovascular effects.
Proportion of participants with demonstrated epinephrine excretion | Days 1-2 of each Arm
  Assays will be performed on participant urine samples to measure the presence of epinephrine metabolites in the form of catecholamines in ng/ml as a measure of cardiovascular effects
Proportion of participants with biomarkers of oxidative stress | Days 1-2 of each Arm
  The proportion of participants with urine samples to measuring oxidative stress-related constituents F2-isoprostane and 11-dehydrothromboxane B2 (dTXB2) in ng/ml will be calculated.
Proportion of participants biomarkers of inflammation | Day 1-2 of each Arm
  The proportion of participants with blood sample results measuring cardiovascular inflammation-related constituents Interleukin 6 (IL-6), Vascular endothelial growth factor (VEGF), and Soluble intercellular adhesion molecule-1 (sICAM-1) in ng/ml will be calculated.

SECONDARY OUTCOMES:
Mean puffs per minute | Day 1 of each Arm
  Vaping topography measures will be obtained from frame-by-frame analysis of high-definition videos during the ad libitum sessions and calculated as mean puffs per minute.
Mean puff duration | Day 1 of each Arm
  Vaping topography measures will be obtained from frame-by-frame analysis of high-definition videos during the ad libitum sessions and calculated as mean seconds per puff.
Mean inter-puff interval | Day 1 of each Arm
  Vaping topography measures will be obtained from frame-by-frame analysis of high-definition videos during the ad libitum sessions and calculated as mean seconds/minutes between puffs.

CONTACTS AND LOCATIONS:
Overall Officials: Gideon St. Helen, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT03839745/Prot_002.pdf
  • Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT03839745/ICF_004.pdf